CLINICAL TRIAL: NCT02437162
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Ustekinumab in the Treatment of Anti-TNF Alpha Naive Subjects With Active Radiographic Axial Spondyloarthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Ustekinumab in the Treatment of Anti-TNFα Naive Participants With Active Radiographic Axial Spondyloarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Neither dose achieved the study's primary or major secondary endpoints. The safety profile was consistent with previous ustekinumab studies.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR107098; CNTO1275AKS3001 (Other: Janssen Research & Development, LLC); 2014-003679-48 (EudraCT Number)
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; Ustekinumab; Golimumab; Stelara
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Ustekinumab; golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo) (Placebo Comparator): Placebo subcutaneous (SC) injection at Weeks 0, 4, and 16. At Week 24 all participants (with the exception of participants who qualified for early escape [EE]) will be re-randomized to receive either ustekinumab 45 or 90 milligram (mg) SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing, with the last administration of study agent at Week 100. Participants who meet EE criteria (less than [<] 10 percent [%] improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and every 4 weeks (q4w) thereafter through Week 52.
  Interventions: Drug: Placebo; Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg; Drug: Golimumab 50 mg
- Group 2 (Ustekinumab 45 mg) (Experimental): Ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by every 12 week dosing, with the last administration of study agent at Week 100. At Week 24, participants will receive placebo SC injection to maintain the blind. Participants who meet EE criteria (<10% improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52.
  Interventions: Drug: Placebo; Drug: Ustekinumab 45 mg; Drug: Golimumab 50 mg
- Group 3 (Ustekinumab 90 mg) (Experimental): Ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 100. At Week 24, participants will receive placebo SC injection to maintain the blind. Participants who meet EE criteria (<10% improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52.
  Interventions: Drug: Placebo; Drug: Ustekinumab 90 mg; Drug: Golimumab 50 mg

INTERVENTIONS:
Drug: Placebo — Participants will receive Placebo subcutaneous (SC) injection at Weeks 0, 4, and 16 in Group 1 and at Week 24 in Group 2 and Group 3.
Drug: Ustekinumab 45 mg — Participants will receive Ustekinumab 45 mg SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing, with the last administration of study agent at Week 100 in Group 1. Participants will start with ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 100 in Group 2.
  Arms: Group 1 (Placebo); Group 2 (Ustekinumab 45 mg)
Drug: Ustekinumab 90 mg — Participants will receive Ustekinumab 90 mg SC injection at Weeks 24 and 28 followed by q12w dosing, with the last administration of study agent at Week 100 in Group 1. Participants will start with ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 100 in Group 3.
  Arms: Group 1 (Placebo); Group 3 (Ustekinumab 90 mg)
Drug: Golimumab 50 mg — Participants who meet EE criteria (less than [<] 10 percent [%] improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and every 4 weeks (q4w) thereafter through Week 52 in Groups 1, 2 and 3.

SUMMARY:
The purpose of this study is to assess the efficacy of ustekinumab, in adult participants with active radiographic axial spondyloarthritis (AxSpA), who are naive to anti-TNF alpha agents, as measured by the reduction in signs and symptoms of radiographic AxSpA.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter (when more than one hospital or medical school team work on a medical research study), randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study. The study consists of 3 phases; Screening (up to 8 weeks), Treatment phase: placebo-controlled (Week 0 to 24) and active treatment (Week 24 to Week 100), and Safety Follow-up (12 weeks after last dose). Participants will be randomly assigned to 1 of 3 treatment groups: placebo, ustekinumab 45 mg and ustekinumab 90 mg. The total duration of study will be up to 112 weeks. Participants will be primarily assessed for Assessment of SpondyloArthritis International Society (ASAS) 40 response at Week 24. Participants' safety will be monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of definite ankylosing spondylitis (AS), as defined by the modified 1984 New York criteria. The radiographic criterion must be confirmed by a central xray reader and at least 1 clinical criterion must be met
* Participants must have symptoms of active disease at screening and at baseline, as evidenced by both a BASDAI score of greater than or equal to (>=4) and a visual analog scale (VAS) score for total back pain of >=4, each on a scale of 0 to 10
* Participants with elevated high sensitivity C-reactive protein (hsCRP) level of >=0.300 milligram per deciliter (mg/dL) at Screening
* If using nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesics for AS, must be on a stable dose for at least 2 weeks prior to the first administration of study agent. If currently not using NSAIDs or other analgesics for AS, must not have received NSAIDs or other analgesics for AS for at least 2 weeks prior to the first administration of the study agent
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test at Week 0 before randomization

Exclusion Criteria:

* Participants who have other inflammatory diseases that might confound the evaluations of benefit from the ustekinumab therapy, including but not limited to, rheumatoid arthritis, systemic lupus erythematosus, or Lyme disease
* Participants who are pregnant, nursing, or planning a pregnancy or fathering a child while enrolled in the study or within 5 months after receiving the last administration of study agent
* Participants who have received any prior biologic therapy, including but not limited to anti-TNF alpha agents, tocilizumab, alefacept, efalizumab, natalizumab, abatacept, anakinra, ustekinumab, tidrakizumab or other anti-interleukin (IL) 23 biologics, brodalumab, secukinumab, ixekizumab, and B-cell depleting therapies
* Participants who have received any systemic immunosuppressives or disease-modifying antirheumatic drugs (DMARDs) other than methotrexate (MTX), sulfasalazine (SSZ), or hydroxychloroquine (HCQ) within 4 weeks prior to first administration of study agent. Medications in these categories include, but are not limited to chloroquine, azathioprine, cyclosporine, mycophenolate mofetil, gold, and penicillamine
* Participant who have received leflunomide within 3 months prior to the first administration of study agent (irrespective of undergoing a drug elimination procedure), or have received leflunomide within 12 months prior to the first administration of study agent and have not undergone a drug elimination procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (57):
- United States (11):
  - Peoria, Arizona
  - St. Petersburg, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Eagan, Minnesota
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Jackson, Tennessee
  - Austin, Texas
  - Mesquite, Texas
  - Seattle, Washington
- Czechia (8):
  - Brno
  - Bruntál
  - Kladno
  - Ostrava
  - Pardubice
  - Prague
  - Uherské Hradiště
  - Zlín
- Poland (5):
  - Bydgoszcz
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
- Russia (16):
  - Chelyabinsk
  - Chita
  - Ivanovo
  - Kemerovo
  - Kirov
  - Kursk
  - Moscow
  - Novosibirsk
  - Orenburg
  - Petrozavodsk
  - Pyatigorsk
  - Saint Petersburg
  - Saratov
  - Stavropol
  - Ufa
  - Ulyanovsk
- South Korea (5):
  - Daegu
  - Daejeon
  - Gwangju
  - Seoul
  - Suwon
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Ukraine (7):
  - Ivano-Frankivsk
  - Kharkiv
  - Lviv
  - Odesa
  - Ternopil
  - Vinnytsia
  - Zaporizhzhya

REFERENCES:
- [Derived] Kavanaugh A, Baraliakos X, Gao S, Chen W, Sweet K, Chakravarty SD, Song Q, Shawi M, Rahman P. Genetic and Molecular Distinctions Between Axial Psoriatic Arthritis and Radiographic Axial Spondyloarthritis: Post Hoc Analyses from Four Phase 3 Clinical Trials. Adv Ther. 2023 May;40(5):2439-2456. doi: 10.1007/s12325-023-02475-4. Epub 2023 Mar 30. PMID 36995469
- [Derived] Deodhar A, Gensler LS, Sieper J, Clark M, Calderon C, Wang Y, Zhou Y, Leu JH, Campbell K, Sweet K, Harrison DD, Hsia EC, van der Heijde D. Three Multicenter, Randomized, Double-Blind, Placebo-Controlled Studies Evaluating the Efficacy and Safety of Ustekinumab in Axial Spondyloarthritis. Arthritis Rheumatol. 2019 Feb;71(2):258-270. doi: 10.1002/art.40728. Epub 2018 Dec 29. PMID 30225992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 347 participants were randomized, and 346 participants were treated (116 participants to placebo, 116 participants to ustekinumab 45 mg, and 114 participants to 90 mg).
Groups:
- Placebo: Participants received placebo subcutaneous (SC) injection at Weeks 0, 4, and 16. At Week 16, participants who met EE criteria were administered open-label golimumab 50 milligram (mg) SC administrations at Week 16 and every 4 weeks (q4w) thereafter through Week 52. At Week 24 all participants (with the exception of participants who qualified for early escape [EE]) were re-randomized to receive either ustekinumab 45 or 90 milligram (mg) SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing through Week 100.
- Ustekinumab 45 mg: Participants received ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by every 12 week dosing through Week 100. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24, participants received placebo SC injection to maintain the blind.
- Ustekinumab 90 mg: Participants received ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing through Week 100. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24, participants received placebo SC injection to maintain the blind.
Period: Overall Study
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Started | 116 | 116 | 115
Treated | 116 | 116 | 114
Early Escape at Week 16 | 26 (Study discontinuation/completion reported under randomization group) | 21 (Study discontinuation/completion reported under randomization group) | 14 (Study discontinuation/completion reported under randomization group)
Cross Over at Week 24 | 87 (Out of 87: crossed over to Ustekinumab 45 mg (n=44) and Ustekinumab 90 mg (n=43)) | 0 | 0
Completed | 9 | 8 | 6
Not Completed | 107 | 108 | 109
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Randomized but not treated | 0 | 0 | 1
Not completed — Study discontinued by Sponsor | 93 | 98 | 97
Not completed — Withdrawal by Subject | 13 | 7 | 9
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least one administration of study agent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | Total
Number analyzed (Participants) | 116 | 116 | 114 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.35) | 39.2 (10.5) | 39.5 (11.32) | 39 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 23 | 14 | 52
  Male | 101 | 93 | 100 | 294
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 1 | 5
  Not Hispanic or Latino | 112 | 116 | 113 | 341
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 30 | 32 | 31 | 93
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 86 | 84 | 82 | 252
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 30 | 32 | 31 | 93
  Black or African American | 0 | 0 | 1 | 1
  Hispanic or Latino | 4 | 0 | 1 | 5
  White Non-Hispanic | 82 | 84 | 81 | 247
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 19 | 14 | 17 | 50
  Ukraine | 19 | 20 | 22 | 61
  United States | 2 | 2 | 1 | 5
  Russia | 32 | 38 | 31 | 101
  Korea, Democratic People'S Republic Of | 9 | 11 | 9 | 29
  Taiwan, Province Of China | 23 | 21 | 23 | 67
  Czech Republic | 12 | 10 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Assessment of Spondyloarthritis International Society (ASAS) 40 Response at Week 24
Description: ASAS 40 defined as improvement from baseline of greater than or equal to (>=) 40 percent (%) and absolute improvement from baseline of at least 2 on 0 to 10 centimeter (cm) scale in at least 3 of following 4 domains: Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation(0 to 10cm;0=none,10=very severe); no worsening at all from baseline in remaining domain. ASAS40 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: The full analysis set (FAS) included all participants who were randomized and received at least one administration of study agent. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received.
Measure: Number; unit: Percentage of participants
Groups:
- Ustekinumab 45 Milligram (mg): Participants received ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by every 12 week dosing through Week 100. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24, participants received placebo SC injection to maintain the blind.
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants | 28.4 | 31.0 | 28.1
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 Milligram (mg); Test type: Superiority; p = 0.669, Cochran-Mantel-Haenszel; Percentage difference = 2.586, 95% CI 2-sided [-9.138 to 14.310]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority; p = 0.913, Cochran-Mantel-Haenszel; Percentage difference = -0.646, 95% CI 2-sided [-12.180 to 10.887]

2. Secondary Outcome: Percentage of Participants Who Achieved an Assessment of Spondyloarthritis International Society (ASAS) 20 Response at Week 24
Description: ASAS 20 defined as improvement from baseline of >= 20% and with an absolute improvement from baseline of 1 on a 0 to 10cm scale in at least 3 of following 4 domains:Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain(0 to 10cm; 0=no pain,10=most severe pain),Bath Ankylosing Spondylitis Functional Index (BASFI) (self-assessment represented as mean(0 to 10 cm; 0=easy to 10=impossible) of 10 questions,8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life, Inflammation (0 to 10cm;0=none,10=very severe);absence of deterioration from baseline(>= 20% and worsening of at least 1 on a 0 to 10 cm scale) in the potential remaining domain. ASAS 20 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: FAS included all participants who were randomized and received at least one administration of study agent. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants | 44.8 | 55.2 | 50.0

3. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50 Percent (%) Improvement From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 24
Description: BASDAI used to measure ankylosing spondylitis (AS) disease severity. Consists of 6 questions: fatigue,spinal pain,arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons, ligaments),morning stiffness(MS) (2 questions:duration, severity). Each question is easy to answer 10cm VAS, 0(none),10(very severe) and for the last question related to morning stiffness duration: 0(0 hours), 10(2 or more hours). In order to give each 5 symptoms equal weight, mean of 2 questions about MS added to total of remaining 4 scores,final BASDAI score(ranging 0-10) is average of overall total score. Higher BASDAI indicates more severe AS symptom. 50% improvement from baseline based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rule(consider non-responder at W20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least one administration of study agent. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants | 27.6 | 25.0 | 25.4

4. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Total Score at Week 24
Description: The BASFI is composed with 10 questions (each question is answered with a visual analogue scale 0-10 cm) to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities of AS participants. Each question is a 10cm VAS with a value between 0 (easy) and 10 (impossible). The final BASFI score is the mean of the 10 scores. The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 10. Higher BASFI score indicates more severe functional limitations of the participant due to AS. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline and Week 24
Population: FAS included all participants who were randomized and received at least one administration of study agent. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 88 | 95 | 99
Units on a scale | -1.85 (2.133) | -2.11 (2.266) | -2.07 (2.502)

5. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score-C Reactive Protein (ASDAS-CRP) Inactive Disease (<1.3) at Week 24
Description: ASDAS includes CRP milligram per liter(mg/L); four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included are total back pain (TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment(PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*TBP) + (0.110*participant global) + (0.073*peripheral pain/swelling) + (0.058* DMS) + (0.579*Ln(CRP+1). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 [normal] to 10 [very severe]) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Inactive disease is defined as an ASDAS score <1.3. ASDAS (CRP) Inactive Disease is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants | 3.4 | 1.7 | 2.6

6. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP) Levels Through Week 24
Description: Change from baseline in hsCRP levels were reported. hsCRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation. Early escape rule was applied(measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: FAS included all participants who were randomized and received at least one administration of study agent. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received. Here 'n' signifies number of participants who were analyzed at each specified timepoint, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Milligrams per deciliter (mg/dL)
  Change at Week 4: number analyzed (Participants) | 115 | 116 | 113
  Change at Week 4 | -0.10 (1.459) | -0.54 (1.488) | -0.74 (1.839)
  Change at Week 8: number analyzed (Participants) | 116 | 115 | 114
  Change at Week 8 | -0.16 (1.478) | -0.59 (1.236) | -0.66 (2.213)
  Change at Week 12: number analyzed (Participants) | 115 | 115 | 112
  Change at Week 12 | -0.18 (1.571) | -0.80 (1.853) | -0.84 (2.262)
  Change at Week 16: number analyzed (Participants) | 115 | 116 | 114
  Change at Week 16 | -0.11 (1.456) | -0.39 (3.166) | -0.86 (2.261)
  Change at Week 20: number analyzed (Participants) | 88 | 93 | 99
  Change at Week 20 | -0.34 (1.450) | -0.73 (1.792) | -0.79 (2.240)
  Change at Week 24: number analyzed (Participants) | 87 | 95 | 98
  Change at Week 24 | -0.41 (1.737) | -0.72 (1.617) | -0.92 (2.274)

7. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) Total Score at Week 16 and 24
Description: Assessment of enthesitis was performed in the following 7 domains: 1) 1st costochondral joint left and right, 2) 7th costochondral joint left and right, 3) posterior superior iliac spine left and right, 4) anterior superior iliac spine left and right, 5) iliac crest left and right, 6) 5th lumbar spinous process and 7) proximal insertion of Achilles tendon left and right. Entheses were scored as either 0 (nontender) or 1 (tender) yielding total MASES ranging from 0 (no tenderness) to 13 (worst possible score; severe tenderness). Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: Population included subset of FAS with enthesitis at baseline. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received. Here 'n' signifies number of participants who were analyzed at each specified timepoint, for each arm.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 87 | 92 | 83
Units on a scale
  Change at Week 16: number analyzed (Participants) | 62 | 59 | 58
  Change at Week 16 | -1.53 (3.347) | -1.47 (3.564) | -1.17 (3.101)
  Change at Week 24: number analyzed (Participants) | 35 | 38 | 44
  Change at Week 24 | -1.66 (3.481) | -1.84 (3.301) | -1.73 (3.060)

8. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 16 and 24
Description: The Bath Ankylosing Spondylitis Metrology Index linear function is a combined index of 5 clinical measurements (performed by the Joint Assessor) which reflect axial mobility in the AS patient. The measurements to assess mobility are: 1)Tragus-to-wall; 2)Modified Schober (lumbar flexion); 3)Cervical rotation angle; 4)Lateral spinal flexion; 5)Intermalleolar distance. The BASMI linear result is the average of the 5 assessments and ranges from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their AS. Early escape rule was applied (measurement value was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 16: number analyzed (Participants) | 114 | 114 | 111
  Change at Week 16 | -0.26 (1.015) | -0.26 (1.044) | -0.17 (0.840)
  Change at Week 24: number analyzed (Participants) | 87 | 92 | 97
  Change at Week 24 | -0.36 (0.943) | -0.37 (0.946) | -0.27 (0.877)

9. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) Score at Week 16 and 24
Description: The ASQoL is a self-administered health-related quality of life (HRQOL) instrument. It consists of 18 items requesting a Yes or No response to questions related to the impact of the disease/condition (including pain) on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. A score of 1 is given to a response of "yes" on each item and all item scores are summed to a total score with a range of 0 to 18. Higher scores indicate worse HRQOL. Early escape rule was applied (measurement value was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 16: number analyzed (Participants) | 114 | 116 | 113
  Change at Week 16 | -2.61 (4.385) | -3.03 (4.416) | -2.93 (3.954)
  Change at Week 24: number analyzed (Participants) | 87 | 94 | 98
  Change at Week 24 | -4.21 (4.441) | -4.48 (4.808) | -4.31 (4.537)

10. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 16 and 24
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worst score) to 52 (best score). Early escape rule was applied (measurement value was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 16: number analyzed (Participants) | 114 | 116 | 113
  Change at Week 16 | 5.71 (9.499) | 5.44 (9.528) | 5.96 (9.325)
  Change at Week 24: number analyzed (Participants) | 87 | 94 | 98
  Change at Week 24 | 8.78 (10.472) | 7.67 (10.348) | 8.59 (10.597)

11. Secondary Outcome: Change From Baseline in Short Form-(SF)-36 Physical Component Summary (PCS) and SF-36 Mental Component Summary (MCS) at Week 16 and 24
Description: The Medical Outcome Study health measure SF-36 questionnaire is a well-validated and widely used quality-of-life instrument. It is a self-administered survey that consists of 8 multi-item scales: The 4 subscales of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and the 4 subscales of the SF-36 comprises the MCS score(vitality, social functioning, role-emotional, and mental health). PCS and MCS are scored from 0 to 100 with higher scores indicating better health (worst value is 0 and best value is 100), which are scored using a norm-based system where linear transformations are performed to transform scores to a mean of 50 and standard deviation of 10. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  SF-36 PCS; change at Week 16: number analyzed (Participants) | 114 | 116 | 114
  SF-36 PCS; change at Week 16 | 4.09 (7.618) | 3.66 (6.172) | 5.17 (6.494)
  SF-36 PCS; change at Week 24: number analyzed (Participants) | 87 | 94 | 98
  SF-36 PCS; change at Week 24 | 7.69 (8.001) | 6.34 (6.198) | 7.20 (7.343)
  SF-36 MCS; change at Week 16: number analyzed (Participants) | 114 | 116 | 114
  SF-36 MCS; change at Week 16 | 4.56 (9.113) | 3.69 (9.690) | 4.06 (9.034)
  SF-36 MCS; change at Week 24: number analyzed (Participants) | 87 | 94 | 98
  SF-36 MCS; change at Week 24 | 5.05 (9.758) | 4.82 (10.841) | 5.46 (8.911)

12. Secondary Outcome: Change From Baseline in BASDAI Inflammation Score Through Week 24
Description: The BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration, severity). Each question is an easy to answer 10 centimeter (cm) visual analog scale (VAS), with 0 being none, and 10 being very severe and for the last question relating to morning stiffness duration: 0(0 hours), 10(2 or more hours). Change from baseline in inflammation was assessed by calculating the average of the Last 2 Questions of the BASDAI Concerning Morning Stiffness. Early escape rule was applied (measurement value was set as missing).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Week 4 | -0.86 (1.650) | -1.09 (1.748) | -1.25 (1.871)
  Week 8: number analyzed (Participants) | 116 | 115 | 114
  Week 8 | -1.45 (1.970) | -1.80 (2.192) | -1.88 (2.160)
  Week 12: number analyzed (Participants) | 116 | 115 | 112
  Week 12 | -1.63 (2.110) | -1.89 (2.143) | -1.88 (2.110)
  Week 16: number analyzed (Participants) | 115 | 116 | 114
  Week 16 | -1.82 (2.221) | -1.98 (2.394) | -1.97 (2.299)
  Week 20: number analyzed (Participants) | 86 | 92 | 98
  Week 20 | -2.48 (2.200) | -2.61 (2.089) | -2.51 (2.429)
  Week 24: number analyzed (Participants) | 88 | 95 | 99
  Week 24 | -2.64 (2.194) | -2.81 (2.257) | -2.74 (2.592)

13. Secondary Outcome: Change From Baseline in Composite and Domain Scores of Medical Outcomes Study Sleep Scale (MOS-SS) at Week 16 and 24
Description: Sleep problems were assessed using the 12-item MOS-SS, a generic instrument designed to assess six dimensions of sleep: Sleep disturbance, Somnolence, Sleep adequacy, Snoring, Awaken short of breath or headache, and Quantity of sleep(QS)/optimal sleep(OS) during the past 4 weeks. The six dimensions were also used to generate the composite Sleep Problems Index (SPI). An increase in score from baseline represents improvement. Sleep disturbance, snoring, somnolence, awaken short of breath, sleep problems index have score ranges from 0(no sleep problems) to 100 (greater sleep problems), negative change indicates improvement. Sleep adequacy scored 0 (least sleep adequacy) to 100 (better sleep adequacy), positive change indicates improvement. Quantity of sleep is scored 0 (less quantity of sleep) to 24 (greater quantity of sleep), positive change indicates improvement. Early escape rule was applied (measurement value was set as missing).
Time Frame: Baseline, Week (W) 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at W16: sleep disturbance: number analyzed (Participants) | 114 | 116 | 113
  Change at W16: sleep disturbance | 3.15 (7.103) | 4.13 (7.815) | 2.79 (6.233)
  Change at W24: sleep disturbance: number analyzed (Participants) | 88 | 94 | 98
  Change at W24: sleep disturbance | 4.57 (7.335) | 5.85 (8.991) | 4.79 (7.232)
  Change at W16: somnolence: number analyzed (Participants) | 114 | 116 | 113
  Change at W16: somnolence | 3.79 (7.996) | 2.06 (7.901) | 2.73 (8.525)
  Change at W24: somnolence: number analyzed (Participants) | 88 | 94 | 98
  Change at W24: somnolence | 4.99 (8.019) | 3.16 (8.612) | 4.52 (9.131)
  Change at W16: sleep adequacy: number analyzed (Participants) | 114 | 116 | 113
  Change at W16: sleep adequacy | 1.78 (7.713) | 1.42 (9.301) | 1.50 (7.851)
  Change-W24: sleep adequacy: number analyzed (Participants) | 88 | 94 | 98
  Change-W24: sleep adequacy | 3.03 (7.245) | 1.75 (9.148) | 3.41 (7.689)
  Change at W16: snoring: number analyzed (Participants) | 114 | 116 | 113
  Change at W16: snoring | 0.47 (7.026) | 1.24 (5.753) | 1.14 (6.520)
  Change at W24: snoring: number analyzed (Participants) | 88 | 94 | 98
  Change at W24: snoring | 0.86 (7.506) | 1.21 (6.715) | 2.64 (7.569)
  Change at W16:awaken short of breath or headache: number analyzed (Participants) | 114 | 116 | 113
  Change at W16:awaken short of breath or headache | 3.93 (12.209) | 3.66 (11.355) | 5.53 (12.602)
  Change-W24:awaken short of breath or headache: number analyzed (Participants) | 88 | 94 | 98
  Change-W24:awaken short of breath or headache | 3.48 (11.179) | 2.76 (11.385) | 3.97 (12.426)
  Change at W16: sleep problems index: number analyzed (Participants) | 114 | 116 | 113
  Change at W16: sleep problems index | 3.72 (7.341) | 3.76 (8.160) | 3.19 (6.695)
  Change at W24:sleep problems index: number analyzed (Participants) | 88 | 94 | 98
  Change at W24:sleep problems index | 5.10 (7.338) | 4.96 (8.794) | 5.16 (7.795)

14. Secondary Outcome: Change From Baseline in Composite and Domain Scores of Medical Outcomes Study Sleep Scale (MOS-SS)-Quantity of Sleep/Optimal Sleep at Week 16 and 24
Description: Sleep problems were assessed using the 12-item MOS-SS, a generic instrument designed to assess six dimensions of sleep: Sleep disturbance, Somnolence, Sleep adequacy, Snoring, Awaken short of breath or headache, QS/OS during past W4. 6 dimensions used to generate composite SPI. Increase in score from baseline represents improvement. Sleep adequacy scored 0 (least sleep adequacy[SA]) to 100 (better SA), positive change indicates improvement. QS is scored 0 (less QS) to 24 (greater QS), positive change indicates improvement. Single-item QS asks participants to estimate average number of hours they slept each night during past 4W (0-24 hours) and transformed into dichotomous OS Score, reported 7 (or 8) hours of sleep considered Optimal. OS is scored Yes if average hours of sleep is in range of 7-8 hours. Early escape rule was applied (measurement value was set as missing).
Time Frame: Baseline, Week (W) 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Hours
  Change-W16: quantity of sleep/optimal sleep: number analyzed (Participants) | 114 | 116 | 113
  Change-W16: quantity of sleep/optimal sleep | 0.15 (0.502) | 0.06 (0.548) | 0.04 (0.557)
  Change-W24: quantity of sleep/optimal sleep: number analyzed (Participants) | 88 | 94 | 98
  Change-W24: quantity of sleep/optimal sleep | 0.16 (0.500) | 0.07 (0.626) | 0.12 (0.579)

15. Secondary Outcome: Percentage of Participants With at Least a 40% Improvement From Baseline in ASAS 40 Components at Week 24
Description: ASAS 40 components included Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe). Percentage of Participants With at least a 40% improvement from baseline in each of the ASAS components was calculated.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 114 | 115 | 113
Percentage of participants
  Patients global assessment | 43.0 | 35.7 | 31.9
  Total back pain | 42.1 | 42.6 | 38.9
  BASFI | 32.5 | 33.0 | 35.4
  Inflammation | 47.4 | 36.5 | 37.2

16. Secondary Outcome: Percentage of Participants Who Achieved at Least 20%, 50%, 70% and 90% Improvement From Baseline in BASDAI Through Week 24
Description: BASDAI used to measure the AS disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration and severity). Each question is an easy to answer cm VAS with 0 being none, and 10 being very severe and for the last question relating to morning stiffness duration: 0(0 hours), 10(2 or more hours). In order to give each of the 5 symptoms equal weight, mean of 2 questions about morning stiffness will be added to total of remaining 4 scores, final BASDAI score (ranging 0-10) is average of overall total score. Higher BASDAI score indicates more severe AS symptom. 20 %,50%, 70%,90% improvement from baseline in BASDAI based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non-responders).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 4 (20% improvement) | 25.9 | 28.4 | 35.1
  Week 8 (20% improvement) | 44.8 | 45.7 | 43.0
  Week 12 (20% improvement) | 47.4 | 45.7 | 41.2
  Week 16 (20% improvement) | 49.1 | 46.6 | 48.2
  Week 20 (20% improvement) | 43.1 | 51.7 | 50.0
  Week 24 (20% improvement) | 47.4 | 55.2 | 51.8
  Week 4 (50% improvement) | 3.4 | 4.3 | 5.3
  Week 8 (50% improvement) | 12.9 | 12.9 | 14.0
  Week 12 (50% improvement) | 19.0 | 12.9 | 14.0
  Week 16 (50% improvement) | 19.8 | 17.2 | 18.4
  Week 20 (50% improvement) | 25.9 | 17.2 | 22.8
  Week 4 (70% improvement) | 0.9 | 0.9 | 1.8
  Week 8 (70% improvement) | 6.9 | 4.3 | 5.3
  Week 12(70 % response) | 6.9 | 6.9 | 7.9
  Week 16(70 % response) | 10.3 | 9.5 | 8.8
  Week 20 (70% improvement) | 11.2 | 6.9 | 10.5
  Week 24 (70% improvement) | 11.2 | 11.2 | 11.4
  Week 4 (90% improvement) | 0 | 0.9 | 0
  Week 8 (90% improvement) | 0.9 | 0 | 1.8
  Week 12 (90% improvement) | 1.7 | 0.9 | 1.8
  Week 16 (90% improvement) | 1.7 | 1.7 | 0.9
  Week 20 (90% improvement) | 2.6 | 0.9 | 1.8
  Week 24 (90% improvement) | 4.3 | 1.7 | 4.4

17. Secondary Outcome: Change From Baseline in BASDAI Total Score Through Week 24
Description: The BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration and severity). Each question is an easy to answer 10 centimeter (cm) visual analog scale (VAS), with 0 being none, and 10 being very severe and for the last question relating to morning stiffness duration: 0(0 hours), 10(2 or more hours). In order to give each of the 5 symptoms equal weight, the mean of the 2 questions about morning stiffness will be added to the total of the remaining 4 scores, and the final BASDAI score (ranging 0-10) is the average of the overall total score. Higher BASDAI score indicates more severe AS symptom. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 4 | -0.83 (1.340) | -0.92 (1.550) | -0.87 (1.632)
  Change at Week 8: number analyzed (Participants) | 116 | 115 | 114
  Change at Week 8 | -1.43 (1.849) | -1.67 (1.984) | -1.49 (2.025)
  Change at Week 12: number analyzed (Participants) | 116 | 115 | 112
  Change at Week 12 | -1.59 (2.073) | -1.64 (2.047) | -1.45 (2.118)
  Change at Week 16: number analyzed (Participants) | 115 | 116 | 114
  Change at Week 16 | -1.67 (2.271) | -1.74 (2.300) | -1.60 (2.276)
  Change at Week 20: number analyzed (Participants) | 86 | 92 | 98
  Change at Week 20 | -2.35 (2.226) | -2.39 (1.922) | -2.20 (2.283)
  Change at Week 24: number analyzed (Participants) | 88 | 95 | 99
  Change at Week 24 | -2.52 (2.262) | -2.56 (2.196) | -2.40 (2.356)

18. Secondary Outcome: Percentage of Participants Who Achieved ASAS 40 Response at Week 4, 8, 12, 16 and 20
Description: ASAS 40 defined as improvement from baseline of greater than or equal to (>=) 40% and with an absolute improvement from baseline of at least 2 on 0 to10cm scale in at least 3 of following 4 domains: Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe); no worsening at all from baseline in remaining domain. ASAS40 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 4 | 7.8 | 6.9 | 8.8
  Week 8 | 14.7 | 18.1 | 19.3
  Week 12 | 19.8 | 14.7 | 18.4
  Week 16 | 22.4 | 21.6 | 22.8
  Week 20 | 22.4 | 22.4 | 28.9

19. Secondary Outcome: Percentage of Participants Who Achieved ASAS 20 Response at Week 4, 8, 12, 16 and 20
Description: ASAS 20 defined as improvement from baseline of greater than or equal to (>=) 20% and with an absolute improvement from baseline of 1 on a 0 to 10 cm scale in at least 3 of following 4 domains: Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe); absence of deterioration (>= 20% and worsening of at least 1 on a 0 to 10 cm scale) from baseline in the potential remaining domain. ASAS20 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 4 | 20.7 | 27.6 | 29.8
  Week 8 | 33.6 | 41.4 | 42.1
  Week 12 | 37.1 | 44.8 | 39.5
  Week 16 | 44.0 | 45.7 | 43.9
  Week 20 | 39.7 | 46.6 | 49.1

20. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis International Society (ASAS) Partial Remission Through Week 24
Description: Low level of disease activity was measured by criteria for ASAS partial remission, defined as a value below 2 on a scale of 0 to 10 cm in each of the 4 ASAS domains: patient's global assessment of disease activity, total back pain, function (BASFI), inflammation. ASAS partial remission response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 4 | 1.7 | 0 | 0.9
  Week 8 | 3.4 | 0.9 | 3.5
  Week 12 | 4.3 | 4.3 | 3.5
  Week 16 | 8.6 | 5.2 | 2.6
  Week 20 | 7.8 | 3.4 | 6.1
  Week 24 | 6.9 | 5.2 | 6.1

21. Secondary Outcome: Percentage of Participants Who Achieved ASAS 5/6 Response at Week 16 and 24
Description: ASAS 5/6 is defined as a >=20% improvement in any 5 of the 6 domains of pain (VAS 0 to 10), patient global (VAS 0 to 10), function (BASFI score), morning stiffness (from BASDAI), hsCRP, and spine mobility (lumbar side flexion). ASAS 5/6 response is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 16 and 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 16 | 23.3 | 29.3 | 26.3
  Week 24 | 30.2 | 35.3 | 33.3

22. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score ASDAS (CRP) Total Score Through Week 24
Description: ASDAS includes CRP mg/L; 4 additional self-reported items (rated 0-10cm VAS or 0-10 numerical rating scale [NRS]) included are total back pain (TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment (PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*TBP)+(0.110*PGA) + (0.073*peripheral pain(PP)/swelling)+(0.058* duration of morning stiffness)+(0.579*Ln(CRP+1)). The disease activity, TBP, and PP/swelling on a NRS(0[normal]-10[very severe]and DMS on NRS(0 to 10, 0 being none and 10 representing a duration=>2 hours). The scores were categorized as: inactive disease (< 1.3), moderate (1.3 - < 2.1), high (2.1 - 3.5) and very high disease activity (> 3.5). The calculated score can be from 0 to no defined upper limit. A negative number indicates a reduction in the score which indicates decrease in disease activity. Early escape rule was applied (measurement value was set as missing).
Time Frame: Baseline, Week 4, 8, 12 ,16, 20 and 24
Population: FAS included all participants who were randomized and received at least one administration of study agent. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received.Here 'n' signifies number of participants who were analyzed at each specified timepoint, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 4: number analyzed (Participants) | 113 | 116 | 113
  Change at Week 4 | -0.41 (0.705) | -0.52 (0.616) | -0.55 (0.673)
  Change at Week 8: number analyzed (Participants) | 114 | 115 | 114
  Change at Week 8 | -0.62 (0.881) | -0.80 (0.764) | -0.75 (0.875)
  Change at Week 12: number analyzed (Participants) | 113 | 114 | 112
  Change at Week 12 | -0.66 (0.957) | -0.87 (0.800) | -0.76 (0.881)
  Change at Week 16: number analyzed (Participants) | 113 | 116 | 114
  Change at Week 16 | -0.67 (1.044) | -0.85 (0.972) | -0.80 (0.926)
  Change at Week 20: number analyzed (Participants) | 84 | 92 | 98
  Change at Week 20 | -1.00 (1.033) | -1.13 (0.844) | -1.01 (0.982)
  Change at Week 24: number analyzed (Participants) | 85 | 95 | 98
  Change at Week 24 | -1.10 (1.088) | -1.19 (0.985) | -1.12 (1.005)

23. Secondary Outcome: Percentage of Participants Who Achieved ASDAS (CRP) Inactive Disease (<1.3) at Week 4, 8, 12, 16 and 20
Description: ASDAS includes CRP mg/L; four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included are total back pain (TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment (PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*total back pain) + (0.110*participant global) + (0.073*peripheral pain/swelling) + (0.058* duration of morning stiffness) + (0.579*Ln(CRP+1)). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Inactive disease is defined as an ASDAS score <1.3. ASDAS (CRP) Inactive Disease is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non- responders).
Time Frame: Week 4, 8, 12, 16, and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 4 | 0.9 | 0 | 0
  Week 8 | 0.9 | 0.9 | 2.6
  Week 12 | 1.7 | 0.9 | 0.9
  Week 16 | 1.7 | 1.7 | 2.6
  Week 20 | 4.3 | 0.9 | 2.6

24. Secondary Outcome: Percentage of Participants With ASDAS (CRP) Major Improvement (Decrease >=2.0) Through Week 24
Description: ASDAS includes CRP mg/L; four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included are total back pain (TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment (PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*TBP) + (0.110*participant global) + (0.073*peripheral pain/swelling) + (0.058* DMS) + (0.579*Ln(CRP+1)). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Major improvement in ASDAS is defined as a decrease from baseline >=2.0. ASDAS (CRP) major improvement (decrease >=2.0) is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non- responders).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 4 | 2.6 | 3.4 | 3.5
  Week 8 | 6.9 | 8.6 | 12.3
  Week 12 | 8.6 | 9.5 | 12.3
  Week 16 | 10.3 | 13.8 | 14.0
  Week 20 | 7.8 | 15.5 | 10.5
  Week 24 | 13.8 | 16.4 | 14.9

25. Secondary Outcome: Percentage of Participants Who Achieved ASDAS (CRP) Clinically Important Improvement (Decrease >=1.1) Through Week 24
Description: ASDAS includes CRP mg/L; four additional self-reported items (rated on 0-10cm VAS or 0-10 NRS) included are TBP, duration of DMS, peripheral pain/swelling and patient global assessment (PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*TBP) + (0.110*participant global) + (0.073*peripheral pain/swelling) + (0.058*DMS) + (0.579*Ln(CRP+1)). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Clinically important improvement in ASDAS is defined as a decrease from baseline >=1.1. ASDAS (CRP) clinical important improvement (decrease >=1.1) is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non- responders).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Percentage of participants
  Week 4 | 16.4 | 13.8 | 17.5
  Week 8 | 26.7 | 31.0 | 30.7
  Week 12 | 28.4 | 37.9 | 28.1
  Week 16 | 32.8 | 35.3 | 28.1
  Week 20 | 29.3 | 31.9 | 37.7
  Week 24 | 37.9 | 40.5 | 37.7

26. Secondary Outcome: Change From Baseline in BASFI at Week 4, 8, 12, 16 and 20
Description: as for outcome 4
Time Frame: Baseline, Week 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 4 | -0.77 (1.635) | -0.80 (1.359) | -0.90 (1.524)
  Change at Week 8: number analyzed (Participants) | 116 | 115 | 114
  Change at Week 8 | -1.13 (1.841) | -1.29 (1.904) | -1.29 (1.841)
  Change at Week 12: number analyzed (Participants) | 116 | 115 | 112
  Change at Week 12 | -1.09 (2.015) | -1.22 (1.854) | -1.34 (2.001)
  Change at Week 16: number analyzed (Participants) | 115 | 116 | 114
  Change at Week 16 | -1.08 (2.179) | -1.35 (2.113) | -1.43 (2.125)
  Change at Week 20: number analyzed (Participants) | 86 | 92 | 98
  Change at Week 20 | -1.71 (2.160) | -1.94 (1.946) | -2.01 (2.291)

27. Secondary Outcome: Change From Baseline in Chest Expansion at Week 16 and 24
Description: Chest expansion is the difference, in centimeter (cm), between the circumference of the chest in maximal inspiration and maximal expiration. It is measured at the level of the fourth intercostal space in males, and just below the breasts in females. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeter(cm)
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
centimeter(cm)
  Change at Week 16: number analyzed (Participants) | 114 | 113 | 111
  Change at Week 16 | 0.43 (7.899) | 0.20 (2.209) | -0.02 (2.240)
  Change at Week 24: number analyzed (Participants) | 87 | 92 | 97
  Change at Week 24 | -0.16 (2.370) | 0.32 (1.939) | -0.21 (2.232)

28. Secondary Outcome: Change From Baseline in Total Back Pain (TBP) and Night Back Pain (NBP) Through Week 24
Description: The total back pain and nighttime back pain was measured on a VAS (0 to 10 cm; 0 = no pain, 10 = most severe pain). Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
centimeter
  Change at Week 4: TBP | -1.13 (2.019) | -1.15 (1.911) | -1.52 (1.895)
  Change at Week 4: NBP | -1.05 (2.270) | -1.25 (1.835) | -1.19 (2.082)
  Change at Week 8: TBP: number analyzed (Participants) | 116 | 115 | 114
  Change at Week 8: TBP | -1.80 (2.190) | -1.78 (2.294) | -2.20 (2.243)
  Change at Week 8: NBP: number analyzed (Participants) | 116 | 115 | 114
  Change at Week 8: NBP | -1.69 (2.264) | -1.85 (2.122) | -2.01 (2.517)
  Change at Week 12: TBP: number analyzed (Participants) | 116 | 115 | 112
  Change at Week 12: TBP | -1.81 (2.295) | -1.70 (2.218) | -1.84 (2.288)
  Change at Week 12: NBP: number analyzed (Participants) | 116 | 115 | 112
  Change at Week 12: NBP | -1.61 (2.342) | -1.79 (2.127) | -1.76 (2.554)
  Change at Week 16: TBP | -1.80 (2.374) | -1.87 (2.465) | -2.07 (2.387)
  Change at Week 16: NBP: number analyzed (Participants) | 115 | 116 | 114
  Change at Week 16: NBP | -1.76 (2.506) | -2.02 (2.541) | -2.05 (2.606)
  Change at Week 20: TBP: number analyzed (Participants) | 86 | 92 | 98
  Change at Week 20: TBP | -2.73 (2.456) | -2.74 (2.088) | -2.69 (2.414)
  Change at Week 20: NBP: number analyzed (Participants) | 86 | 92 | 98
  Change at Week 20: NBP | -2.67 (2.602) | -2.73 (2.246) | -2.83 (2.804)
  Change at Week 24: TBP: number analyzed (Participants) | 88 | 95 | 99
  Change at Week 24: TBP | -2.80 (2.528) | -2.90 (2.389) | -2.77 (2.511)
  Change at Week 24: NBP: number analyzed (Participants) | 88 | 94 | 99
  Change at Week 24: NBP | -2.75 (2.597) | -2.79 (2.367) | -2.68 (2.960)

29. Secondary Outcome: Change From Baseline in Patients Global Assessment of Disease Activity Through Week 24
Description: Participants assessed their disease activity using a 10 cm visual analog scale, with responses ranging from 0 (very well) to 10 (very poor). Early escape rule was applied (The measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 4 | -0.99 (1.727) | -1.01 (1.677) | -1.21 (1.645)
  Change at Week 8: number analyzed (Participants) | 116 | 115 | 114
  Change at Week 8 | -1.48 (2.086) | -1.60 (2.039) | -1.70 (2.096)
  Change at Week 12: number analyzed (Participants) | 116 | 115 | 112
  Change at Week 12 | -1.52 (2.043) | -1.53 (2.100) | -1.77 (2.088)
  Change at Week 16: number analyzed (Participants) | 115 | 116 | 114
  Change at Week 16 | -1.64 (2.259) | -1.73 (2.564) | -1.77 (2.293)
  Change at Week 20: number analyzed (Participants) | 86 | 92 | 98
  Change at Week 20 | -2.10 (2.272) | -2.17 (2.225) | -2.36 (2.283)
  Change at Week 24: number analyzed (Participants) | 88 | 95 | 99
  Change at Week 24 | -2.37 (2.298) | -2.55 (2.664) | -2.50 (2.379)

30. Secondary Outcome: Change From Baseline in European Quality of Life 5 Dimension (EQ-5D) Visual Analog Scale (VAS) Score at Week 16 and 24
Description: The EQ-5D questionnaire is a brief, generic health-related quality of life assessment (HRQOL) that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health). Lower scores indicate worsening. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Change at Week 16: number analyzed (Participants) | 114 | 116 | 113
  Change at Week 16 | 11.49 (20.328) | 11.26 (23.588) | 13.36 (22.110)
  Change at Week 24: number analyzed (Participants) | 87 | 94 | 98
  Change at Week 24 | 17.57 (20.251) | 13.90 (26.132) | 16.80 (22.181)

31. Secondary Outcome: Change From Baseline in EQ-5D Index Score at Week 16 and 24
Description: The EuroQol-5 is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing death. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
Units on a scale
  Week 16: number analyzed (Participants) | 114 | 116 | 113
  Week 16 | 0.08 (0.138) | 0.09 (0.154) | 0.10 (0.139)
  Week 24: number analyzed (Participants) | 87 | 94 | 98
  Week 24 | 0.12 (0.137) | 0.12 (0.168) | 0.13 (0.153)

32. Secondary Outcome: Change From Baseline in Berlin Magnetic Resonance Imaging (MRI) Spine Score at Week 24
Description: The study used MRI with fat-saturating techniques such as short tau inversion recovery (STIR) to look for the presence of bone marrow edema. The Berlin modification of Ankylosing Spondylitis spine MRI score for activity (ASspiMRI-a) scoring technique assesses inflammation in each of the 23 disc vertebral units (DVU), capturing edema and erosion. Scores for each DVU range from 0-3 (0=normal; 1=minor bone marrow edema [less than or equal to 25% of DVU; 3=severe bone marrow edema (more that 50% of DVU)]. The composite score ranges from 0 to 69, with higher scores indicating more severe inflammation.
Time Frame: Baseline and Week 24
Population: Population included subset of FAS with participants who did not meet early escape criteria and have both baseline and Week 24 MRI assessments.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 23 | 18 | 26
Units on a scale | -0.48 (2.053) | -0.58 (2.343) | -1.15 (2.323)

33. Secondary Outcome: Change From Baseline in Percent Work Time Missed Due to AS (Assessed by Work Productivity and Activity Impairment Questionnaire - Specific Health Problem [WPAI-SHP]) Through Week 24
Description: The WPAI-SHP is a 6-item questionnaire used to assess the degree to which a specified health problem (here "AS") affected work attendance, work productivity and productivity in non-work regular activities. Patients are asked to consider the past 7 days prior to each questionnaire day. The questionnaire asks: current employment status, hours worked, hours missed from work for any reason other than AS, hours missed from work due to AS, degree to which AS affected work productivity, and degree to a which AS affected non-work regular activities. Four component scores were then calculated: percent work time missed due to AS; percent impairment while working due to AS, percent overall work impairment due to AS, and percent non-work activity impairment due to AS. The computed percentage range for each sub-scale was from 0-100, with higher numbers indicating greater impairment and less productivity. change from baseline in percent work time missed due to AS for each study arm are reported.
Time Frame: Baseline, Week 16 and 24
Population: FAS included participants who were randomized and received at least one administration of study agent. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received. Here 'n' signifies number of participants who were analyzed at each specified timepoint, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
units on a scale
  Change at Week 16: number analyzed (Participants) | 67 | 67 | 70
  Change at Week 16 | -3.72 (26.092) | -2.05 (26.625) | -2.06 (26.486)
  Change at Week 24: number analyzed (Participants) | 55 | 56 | 62
  Change at Week 24 | -7.37 (16.925) | -4.38 (22.562) | -7.07 (22.081)

34. Secondary Outcome: Change From Baseline in Percent Impairment While Working Due to AS (Assessed by WPAI-SHP) Through Week 24
Description: WPAI-SHP is 6-item questionnaire used to assess the degree to which a specified health problem ("AS") affected work attendance, work productivity and productivity in non-work regular activities. Patients are asked to consider the past 7 days prior to each questionnaire day. The questionnaire asks: current employment status, hours worked, hours missed from work for any reason other than AS, hours missed from work due to AS, degree to which AS affected work productivity, and degree to a which AS affected non-work regular activities. Four component scores were then calculated: percent work time missed due to AS; percent impairment while working due to AS, percent overall work impairment due to AS, and percent non-work activity impairment due to AS. The computed percentage range for each sub-scale was from 0-100, with higher numbers indicating greater impairment and less productivity. change from baseline in percent impairment while working due to AS for each study arm are reported.
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
units on a scale
  Change at Week 16: number analyzed (Participants) | 67 | 67 | 70
  Change at Week 16 | -16.87 (25.359) | -5.97 (21.607) | -17.57 (20.032)
  Change at Week 24: number analyzed (Participants) | 55 | 56 | 62
  Change at Week 24 | -22.00 (21.892) | -13.57 (22.758) | -19.68 (22.973)

35. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment Due to AS (Assessed by WPAI-SHP) Through Week 24
Description: WPAI-SHP is 6-item questionnaire used to assess the degree to which a specified health problem (AS) affected work attendance, work productivity and productivity in non-work regular activities. Patients are asked to consider the past 7 days prior to each questionnaire day. Questionnaire asks: current employment status, hours worked, hours missed from work for any reason other than AS, hours missed from work due to AS, degree to which AS affected work productivity, and degree to a which AS affected non-work regular activities. Four component scores were then calculated: percent work time missed due to AS; percent impairment while working due to AS, percent overall work impairment due to AS, percent non-work activity impairment due to AS. The computed percentage range for each sub-scale was from 0-100, with higher numbers indicating greater impairment and less productivity. change from baseline in percent overall work impairment due to AS for each study arm are reported.
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
units on a scale
  Change at Week 16: number analyzed (Participants) | 67 | 67 | 70
  Change at Week 16 | -16.03 (26.281) | -6.64 (23.976) | -17.48 (20.811)
  Change at Week 24: number analyzed (Participants) | 55 | 56 | 62
  Change at Week 24 | -21.98 (21.042) | -14.64 (24.300) | -20.54 (24.271)

36. Secondary Outcome: Change From Baseline in Percent Non-work Activity Impairment Due to AS (Assessed by WPAI-SHP) Through Week 24
Description: WPAI-SHP is6-item questionnaire used to assess the degree to which a specified health problem (AS) affected work attendance, work productivity and productivity in non-work regular activities. Patients are asked to consider the past 7 days prior to each questionnaire day. The questionnaire asks: current employment status, hours worked, hours missed from work for any reason other than AS, hours missed from work due to AS, degree to which AS affected work productivity, and degree to a which AS affected non-work regular activities. Four component scores were then calculated: percent work time missed due to AS; percent impairment while working due to AS, percent overall work impairment due to AS, and percent non-work activity impairment due to AS. The computed percentage range for each sub-scale was from 0-100, with higher numbers indicating greater impairment and less productivity. change from baseline in percent non-work activity impairment due to AS for each study arm are reported.
Time Frame: Baseline, Week 16 and 24
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ustekinumab 45 Milligram (mg) | Ustekinumab 90 mg
Number analyzed (Participants) | 116 | 116 | 114
units on a scale
  Change at Week 16: number analyzed (Participants) | 114 | 116 | 113
  Change at Week 16 | -14.74 (23.013) | -13.45 (21.833) | -17.52 (22.101)
  Change at Week 24: number analyzed (Participants) | 87 | 94 | 98
  Change at Week 24 | -21.72 (23.288) | -21.49 (23.825) | -21.73 (22.339)

ADVERSE EVENTS:
Time Frame: Approximately 2 years
Description: The safety analysis set included all participants who received at least 1 (partial or complete) administration of study agent, i.e., the treated population. Adverse events were reported according to the treatment they actually received, regardless of the treatments they are randomized to.
Groups:
- Placebo Only: Participants received placebo subcutaneous (SC) injection at Weeks 0, 4, and 16. At Week 16, participants who met EE criteria were administered open-label golimumab 50 milligram (mg) SC administrations at Week 16 and every 4 weeks (q4w) thereafter through Week 52. At Week 24 all participants (with the exception of participants who qualified for early escape [EE]) were re-randomized to receive either ustekinumab 45 or 90 milligram (mg) SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing through Week 100.
- Placebo to Golimumab: Participants randomized to placebo SC who met early escape criteria and received golimumab 50 mg from Week 16; adverse events are counted from early escape onward.
- Placebo to Ustekinumab 45mg: Participants randomized to placebo SC and then rerandomized to receive ustekinumab 45 mg at Week 24; adverse events are counted from crossover onward.
- Placebo to Ustekinumab 90mg: Participants randomized to placebo SC and then rerandomized to receive ustekinumab 90 mg at Week 24; adverse events are counted from crossover onward.
- Ustekinumab 45 mg Only: Participants received ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by every 12 week dosing through Week 100. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52.
- Ustekinumab 45mg to Golimumab: Participants randomized to ustekinumab 45 mg SC who met early escape criteria and received golimumab 50 mg from Week 16; adverse events are counted from early escape onward.
- Ustekinumab 90 mg Only: Participants received ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing through Week 100. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52.
- Ustekinumab 90mg to Golimumab: Participants randomized to ustekinumab 90 mg SC who met early escape criteria and received golimumab 50 mg from Week 16; adverse events are counted from early escape onward.
Arm/Group | Placebo Only | Placebo to Golimumab | Placebo to Ustekinumab 45mg | Placebo to Ustekinumab 90mg | Ustekinumab 45 mg Only | Ustekinumab 45mg to Golimumab | Ustekinumab 90 mg Only | Ustekinumab 90mg to Golimumab
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/26 | 0/44 | 0/43 | 0/116 | 1/21 | 0/114 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/116 | 0/26 | 2/44 | 2/43 | 3/116 | 3/21 | 2/114 | 0/14
Other Adverse Events (participants affected / at risk) | 15/116 | 4/26 | 3/44 | 0/43 | 24/116 | 7/21 | 26/114 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Only (N=116) | Placebo to Golimumab (N=26) | Placebo to Ustekinumab 45mg (N=44) | Placebo to Ustekinumab 90mg (N=43) | Ustekinumab 45 mg Only (N=116) | Ustekinumab 45mg to Golimumab (N=21) | Ustekinumab 90 mg Only (N=114) | Ustekinumab 90mg to Golimumab (N=14)
Ocular Hypertension (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA Version 20.0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
Appendicitis (Infections and infestations) | 0 (0) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA Version 20.0
Back Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA Version 20.0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA Version 20.0,
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA Version 20.0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA Version 20.0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA Version 20.0
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA Version 20.0
Facial Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA Version 20.0
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA Version 20.0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Only (N=116) | Placebo to Golimumab (N=26) | Placebo to Ustekinumab 45mg (N=44) | Placebo to Ustekinumab 90mg (N=43) | Ustekinumab 45 mg Only (N=116) | Ustekinumab 45mg to Golimumab (N=21) | Ustekinumab 90 mg Only (N=114) | Ustekinumab 90mg to Golimumab (N=14)
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 — MedDRA Version 20.0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 — MedDRA Version 20.0
Respiratory Tract Infection Viral (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 6 | 0 — MedDRA Version 20.0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 0 | 0 | 3 | 2 | 4 | 0 — MedDRA Version 20.0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 | 1 | 1 | 0 | 9 | 2 | 11 | 0 — MedDRA Version 20.0
Alanine Aminotransferase Increased (Investigations) | 6 | 2 | 1 | 0 | 8 | 2 | 6 | 0 — MedDRA Version 20.0
Aspartate Aminotransferase Increased (Investigations) | 3 | 2 | 0 | 0 | 8 | 3 | 3 | 0 — MedDRA Version 20.0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 — MedDRA Version 20.0
Ankylosing Spondylitis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA Version 20.0
Fasciitis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA Version 20.0

LIMITATIONS AND CAVEATS:
The study was terminated since neither dose achieved the study's primary or major secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT02437162/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT02437162/SAP_001.pdf